CLINICAL TRIAL: NCT05818631
Title: Determine the Validity as a Diagnostic Test of the Transrectal Prostate Biopsy With Cognitive Fusion Through Biparametric Magnetic Resonance in the Detection of Non-palpabe Prostate Cancer
Brief Title: Cognitive Fusion Prostate Biopsy With Biparametric Magnetic Resonance in the Detection of Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: José Joaquín Mira (Other)
Responsible Party: Sponsor-Investigator, José Joaquín Mira, Director, Universidad Miguel Hernandez de Elche
Organization: Universidad Miguel Hernandez de Elche (Other)
Other Study IDs: Prostate MRI FAST protocol
Record Dates: First submitted 2023-04-04; First posted 2023-04-19 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer; Prostate Cancer Diagnosis
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRI +: PI-RADS 3-5
  Interventions: Diagnostic Test: fusion cognitive prostate biopsy
- MRI -: PI-RADS 1-2

INTERVENTIONS:
Diagnostic Test: fusion cognitive prostate biopsy — A standard transrectal prostatic biopsy will be performed to both groups. To the group with suspicious lesions in the MRI (PI-RADS 3-5), an added directed cognitive fusion biopsy will be performed.
  Other Names: directed prostate biopsy
  Groups: MRI +

SUMMARY:
The goal of this prospective observational study is to evaluate the diagnostic precision of the Biparametric Magnetic Resonance Imaging (bpMRI) in the detection of clinically significant prostate cancer (PCa) in patients with biochemical suspicion of prostate cancer with PSA (Prostate Specific Antigen) > 4 ng/mL and a normal digital rectal examination and without a biopsy previous to the MRI. Secondary aims are:

* Determine the validity as a diagnostic test of the first directed transrectal prostatic biopsy (cognitive fusion) versus systematic biopsy of 12 cylinders in patients with suspicious lesions in the bpMRI.
* Develop a predictive nomogram that permits the reduction of the number of prostatic biopsies performed to patients with a low suspicion of prostate cancer in the bpMRI.

DETAILED DESCRIPTION:
In Spain, PCa is the most common cancer independently from gender and the third cause of death in man, below lung and colorectal cancer. Incidence and mortality increase progressively as age increases, hence, due to an older population, this is an outstanding sociosanitary concern.

PCa generally is asymptomatic, diagnosis is based on prostate biopsy in man with an elevated Prostate Specific Antigen (PSA) in blood test and/or a pathologic digital rectal examination.

Multiparametric Magnetic Resonance Imaging (MRImp) plays an important role in the diagnosis. It allows the visualization of the tumor, it values its agresitivity with a scale named "Prostate Imaging-Reporting and Data System" (PI-RADS v2 scale), and permits a directed biopsy to the suspicious lesion.

This tecnique is expensive and very uncomfortable for the patient due its duration (40 minutes) and because it uses intravenous (iv) contrast. Due to these reasons, it is difficult to assume by the sanitary system to perform this technique to every patient with PCa suspicion.

Biparametric MRI emerges as an alternative with a new protocol, performed with less image sequences (T2 and diffusion), cheaper, lasting less (just 15 minutes), and without the administration of iv contrast. Thus, this technique is more assumable by a public sanitary system.

ELIGIBILITY:
Inclusion Criteria:

* Male patients between 18 and 80 years
* BpMRI performed in a 3 months period before the prostatic biopsy
* First transrectal prostatic biopsy
* PSA > 4 ng/mL and < 20 ng/mL
* Patients acceptance to participate in the study signing a written specific informed consent

Exclusion Criteria:

* Not having all the inclusion criteria described
* Suspicious digital rectal examination of prostate cancer
* Previous urinary tract infection in the last six months, acute urinary retention or being a chronic carrier of bladder catheter
* Previous prostatic surgery in any of its variants
* Concomitant treatment with Luteinizing hormone-releasing hormone (LHRH) analogue, antiandrogens or 5-alfa-reductase inhibitors

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed in the 17th department of the Valencian Community (San Juan de Alicante's Department).
  Main patients are those that visit the consultation room in the Urological department of the Hospital Universitario San Juan de Alicante.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic precision of Biparametric Magnetic Resonance Imaging: consecutive validation of two diagnostic tests for obtaining sensitivity, specificity, positive predictive value and negative predictive value of the biparametric magnetic resonance imaging | 1 hour
  evaluate the diagnostic precision of the Biparametric Magnetic Resonance Imaging (bpMRI) in the detection of clinically significant prostate cancer in patients with biochemical suspicion of prostate cancer (Prostate Specific Antigen in blood test > 4 ng/mL) with a normal digital rectal examination and without a biopsy previous to the MRI

SECONDARY OUTCOMES:
Validity of first directed transrectal prostatic biopsy: consecutive validation of two diagnostic tests for obtaining sensitivity, specificity, positive predictive value and negative predictive value of the biparametric magnetic resonance imaging | 1 hour
  Determine the validity as a diagnostic test of the first directed transrectal prostatic biopsy (cognitive fusion) versus systematic biopsy of 12 cylinders in patients with suspicious lesions in the bpMRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Miguel Hernández de Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided